CLINICAL TRIAL: NCT00277563
Title: Short and Long Term Exposure to Unique, Time-Varying Pulsed Electro-Magnetic Fields in Refractory Carpal Tunnel Syndrome (Cts): A Randomized, Placebo-Controlled Trial With Secondary Bayesian Modification
Brief Title: Short and Long Term Exposure to Unique, Time-Varying Pulsed Electro-Magnetic Fields in Refractory Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weintraub, Michael I., MD, FACP, FAAN (Individual)
Collaborators: Dr. Steven P. Cole, PhD. Statistician (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-Weintraub
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Refractory Carpal Tunnel Syndrome; Neurpathic Pain; Neuromodulaton
Keywords: Carpal Tunnel Syndrome; Neuropathic Pain; Neuromodulation; PEMF; Magnetic Field Therapy; Magnetotherapy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Neuralgia

INTERVENTIONS:
Device: reduction of pain scores by magnetic energy

SUMMARY:
Pulsed electromagnetic fields (PEMF) have been approved by FDA and are utilized currently in treating non-union fractures, neurogenic bladder and musculoskeletal pains. Based on 2 prior pilot studies (open label) demonstrating reduction in neuropathic pain from carpal tunnel syndrome we decided to perform a placebo-controlled trial, randomized for 2 months utilizing a wrist PEMF device attached by Velcro for 4 hours/day.

DETAILED DESCRIPTION:
INTRODUCTION:

Entrapment of the median nerve at the wrist is the most common cause of sensory and motor disturbance in the hands and can be progressively disabling.1,2 Complex mechanisms of compression and ischemia exist that adversely influence the large A myelinated fibers and small unmyelinated nociceptive C fibers. From a pathophysiological standpoint, neuropathic pain (numbness, tingling and burning, NP) is believed secondary to ectopic firing of nociceptive afferent unmyelinated C-fiber axons that are undergoing degeneration.3 Microneurography has confirmed that dysregulated expression of sodium and calcium channels, which accumulate at site of injury, are responsible for ectopic depolarization.3,4,53,54 When conventional therapy of splinting and pharmacotherapy fail, surgical decompression has been offered for moderate-severe cases. While usually successful, it is associated with significant complications, limitations and costs.5,6,7 Thus, the search for reliable and new therapeutic strategies is appealing.

Substantial evidence exists that time-varying magnetic fields produce biological effects by safely inducing extremely low-frequency (ELF) small electrical eddy currents within the tissues that can depolarize, repolarize and hyperpolarize neurons.8,9,10,11,12

Prior pilot data using static13 and pulsed magnetic fields (PEMF)14,15 directed to the carpal tunnel region significantly reduced NP. Since a new, novel device became commercially available that produced a combination of static and time-varying magnetic fields simultaneously, it was hypothesized that this energy could be directed into the wrists and potentially influence not only NP scores, but also modulate neuronal distal latencies (neurotransmission).

DEVICE:

DESCRIPTION: (FIGURE 1) This patented device (Biaxial Super Mini [Mx2R] by Nikken, Inc.) measures 2" in diameter and 1" in height and is worn with a Velcro strap similar to a wristwatch. It is noiseless and nonthermal. Its main component is a spherical permanent magnet, 1150G, 3/8" in diameter that rotates in two perpendicular directions simultaneously producing biaxial magnetic rotation (MX2R) and oscillating polarities up to 1,200 rpm-20 times per second. It is driven by a 2 V DC micro-motor which is shielded one inch away and produces a negligible back EMF. The device is powered by three ¼ AAA rechargeable NiMH (Nickel Metal Hydride) batteries

Randomized double blind placebo-controlled device with primary parameters of pain and sleep interupption scores, NPS scale and secondary parameters of neurological exam changes, nerve conduction latencies of median nerve, dynamometry, finger gauge pressures, CPT and PGIC were compared at baseline and end of two months. Patients were given a free "active" device gratis at end of study.

ELIGIBILITY:
Inclusion Criteria:

* Intractable neuropathic pain in median nerve innervated hand for at least 3 months;
* Abnormal neurological examination compatible with diagnosis of CTS

Exclusion Criteria:

* Post-surgical failures,
* Pregnancy,
* Pts with pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-06; Study Completion 2005-07

PRIMARY OUTCOMES:
VAS Pain scores 0-10 (leikert scale)
VAS Sleep interrupption 0-10
Neuropathic Pain scale (NPS)

SECONDARY OUTCOMES:
Neurological Exam
Median nerve distal latencies (CMAP/SNAP)
Hand help Dynamometry and Finger gauge pressures
CPT (Neurometer)
PGIC

CONTACTS AND LOCATIONS:
Overall Officials: Steven P. Cole, PhD, Study Chair — Statistician
Locations (1):
- Michael I. Weintraub MD, PC, Briarcliff, New York, United States

REFERENCES:
- [Derived] Weintraub MI, Cole SP. A randomized controlled trial of the effects of a combination of static and dynamic magnetic fields on carpal tunnel syndrome. Pain Med. 2008 Jul-Aug;9(5):493-504. doi: 10.1111/j.1526-4637.2007.00324.x. PMID 18777606